CLINICAL TRIAL: NCT00691119
Title: A Feasibility Study of Relaxation and Visualization Therapy for Breast Cancer Patients
Brief Title: Relaxation and Visualization Therapy for Breast Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate recruitment
Sponsor: National University of Natural Medicine (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Heather Zwickey, Dean of Research, National University of Natural Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00003439
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; radiation; Relaxation and Visualization Therapy; relaxation; visualization; RVT; complementary and alternative medicine; CAM; alternative medicine
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Relaxation and Visualization Therapy group
  Interventions: Behavioral: Relaxation and Visualization Therapy
- B (Active Comparator): Health education group
  Interventions: Other: Health education
- C (No Intervention): Control group

INTERVENTIONS:
Behavioral: Relaxation and Visualization Therapy — Twenty minutes of facilitated relaxation and visualization therapy five days a week for six weeks. Self practice of 20 minutes per day for the next six weeks.
  Other Names: RVT
  Arms: A
Other: Health education — Facilitated health education sessions, twenty minutes, five times a week for six weeks.
  Arms: B

SUMMARY:
The purpose of this study is to find out if it is possible to study relaxation and visualization therapy (RVT) with individuals that have breast cancer. We will also look at what effects, the good and bad, RVT has when used with radiation therapy. We are interested in how RVT may relate to energy, quality of life, stress, and the immune system. Relaxation and Visualization therapy will lead participants through a practice of physical relaxation and then a step by step visualization. In this study, participants will be led through an RVT exercise, providing an interactive process. In addition, women will perform solitary RVT exercises at home on weekends. Participants for this study will be drawn from two OHSU physicians' regular patient base. To be sure that we are testing the effects of RVT alone, we will use three groups. The three groups will be RVT, education, and a control. The RVT group will receive RVT with radiation, and the education group will receive breast cancer related health education with radiation. The third group will receive no treatment beyond radiation. This third group is called the control. The entire study will last for approximately twelve weeks. For the first 6 weeks, each participant will be receiving radiation therapy. We will be particularly interested in the effects that RVT may have on energy, quality of life, stress, and the immune system. No experimental drug or device will be used during the study.

DETAILED DESCRIPTION:
The purpose of this study is to find out if it is possible to study relaxation and visualization therapy (RVT) with individuals that have breast cancer. We will also look at what effects, the good and bad, RVT has when used with radiation therapy. We are interested in how RVT may relate to energy, quality of life, stress, and the immune system. Relaxation is a state in which the body slows down, like in sleep or rest. Heart rate decreases, breathing slows and digestion increases. Visualization is an interactive mental process. The participant imagines herself doing a physical activity. This imagination stimulates a measurable physical response. Relaxation and Visualization therapy will lead participants through a practice of physical relaxation and then a step by step visualization. RVT can be performed by an individual alone, or it can be led by a health practitioner. In this study, participants will be led through an RVT exercise, providing an interactive process. In addition, women will perform solitary RVT exercises at home on weekends. Participants for this study will be drawn from two OHSU physicians' regular patient base. Newly diagnosed patients will be offered the opportunity to participate in our Relaxation and Visualization Therapy Study. We want to make sure that the results we see are not due to any other factors. To be sure that we are testing the effects of RVT alone, we will use three groups. The three groups will be RVT, education, and a control. The RVT group will receive RVT with radiation, and the education group will receive breast cancer related health education with radiation. Both test groups will last approximately one hour. The third group will receive no treatment beyond radiation. This third group is called the control. The entire study will last for approximately twelve weeks. For the first 6 weeks, each participant will be receiving radiation therapy. The second 6 weeks will be done mostly at home. We will be particularly interested in the effects that RVT may have on energy, quality of life, stress, and the immune system. To examine this, participants will complete surveys about stress and psychological changes. A dietary assessment will be conducted via interviews. Participants will be asked to recall what foods commonly eaten. A heart monitor will be worn during the educational and visualization activities to monitor any changes in heart rate. Additionally, 5 blood draws will occur during the study, and the total amount of blood drawn will be about 4 tablespoons of blood. No experimental drug or device will be used during the study.

ELIGIBILITY:
Inclusion Criteria:

* women who have been diagnosed with breast cancer and have been referred to radiotherapy at OHSU
* between 45 and 70 years of age

Exclusion Criteria:

* receiving chemotherapy concurrently
* uses tobacco products
* has a fear or aversion to blood draws
* has a history of hypertension
* uses recreational drugs
* drinks more than 3-5 alcoholic beverages per week
* takes any anti-inflammatory medications
* has a current infection or has a compromised immune system

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Establish methodological feasibility for a larger study of RVT for women with breast cancer receiving radiotherapy | Ongoing
Time of onset, length, and severity of fatigue with the Schwartz Cancer Fatigue Scale (SCFS) | Five days a week for six weeks

SECONDARY OUTCOMES:
Radiation Therapy Oncology Group (RTOG) Acute Skin Toxicity scale | Once a week for six weeks
Quality of Life [SF-36] | Once during week 1, week 6 and week 12 of intervention
Perceived Stress Scale | Once during week 1, week 6 and week 12 of intervention
State and Trait Anxiety Inventory[STAI] | Once during week 1, week 6 and week 12 of intervention
Functional Assessment of Cancer Therapy-Breast [FACT-B] | Once during week 1, week 6, and week 12 of intervention
Transformative Change Scale | Once during week 1, week 6, and week 12 of intervention
Diet inquiry | once during week 6 and week 12 of intervention
Heart rate monitoring | Five days a week during six week intervention, once during final week 12 visit
Adverse events | During radiation visits (five times a week for six weeks) with doctor/principal investigator, week 6 and week 12 visit
Immune assessments via blood testing: IL-6, IL-1, IL-ra, IL-4, IL-8, IL-10, TNFalpha, IFNgamma, and CRP | Once every other week for 12 week study period
Neurological assessments via blood testing: serotonin, GABA and norepinephrine | Once every other week for the 12 week study period

CONTACTS AND LOCATIONS:
Overall Officials: Carol Marquez, MD, Principal Investigator — Oregon Health and Science University; Heather Zwickey, PhD, Principal Investigator — Helfgott Research Institute at National College of Natural Medicine
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States